CLINICAL TRIAL: NCT03475485
Title: Clinical Performance of the ID-Cap System, an Ingestion Event Marker, in the Clinical Setting as an Aid to Measure Medication Adherence
Brief Title: ID-Cap System Under Direct Observation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: EtectRX, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Device Feasibility
Other Study IDs: ERX001
Record Dates: First submitted 2018-03-18; First posted 2018-03-23 (Actual); Last update posted 2018-06-11 (Actual); Status verified 2018-06

CONDITIONS: Healthy Volunteers
Keywords: Ingestion event marker; Ingestible sensor; Medication adherence; ID-Cap Medication Adherence Feedback System
MeSH Terms: conditions — Medication Adherence

STUDY DESIGN:
Intervention Model Description: This study is a prospective, blinded, clinical study evaluating the safety and effectiveness of the ID-Cap System under direct observation in the clinical setting. Subjects will ingest a series of active ID capsules containing ingestible sensors and a series of empty placebo capsules that will be randomly administered. The ID-Capsule System's feasibility/ability to properly record actual ingestions (Positive Detection Accuracy) and to not record blank ingestions (Negative Detection Accuracy) will be evaluated.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Capsules are identical in appearance. Only unblinded pharmacy personnel at the study site will be aware of the ingestion allocation of active ID-Capsules or placebo capsules.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- ID-Capsules- Active (Experimental): Randomly-assigned ingestions of ID-Capsules containing ingestible sensors (ID-Capsule- Active) while wearing the ID-Cap Reader (Wearable Sensor) under direct observation
  • Subjects will ingest ID-Capsules containing the ingestible sensor which emits a signal from within the subject's stomach. This signal is detected by the wearable Reader, and the ingestion event is recorded.
  Interventions: Device: ID-Capsule- Active; Device: Wearable Sensor
- ID-Capsules- Inactive (Placebo Comparator): Randomly-assigned ingestions of ID-Capsules containing no ingestible sensors while wearing the ID-Cap Reader under direct observation
  • Subjects will also ingest empty placebo capsules that do not contain ingestible sensors. In the absence of an ingested sensor, no signal is received by the Reader after the capsule is ingested, and the ingestion event is not recorded.
  Interventions: Device: Wearable Sensor; Device: Placebo

INTERVENTIONS:
Device: ID-Capsule- Active — A standard gelatin or HPMC capsule with an embedded ingestible wireless sensor.
  Arms: ID-Capsules- Active
Device: Wearable Sensor — Subjects will wear an ID-Reader
Device: Placebo — A standard gelatin or HPMC capsule without an embedded ingestible wireless sensor.
  Arms: ID-Capsules- Inactive

SUMMARY:
The ID-Cap System is classified as an ingestion event marker (IEM), a Class II medical device. The system is intended to record time-stamped ingestions with the ingestible sensor, ID-Tag which transmits a signal to a wearable device, the ID-Cap Reader. In this study, 36 subjects will ingest capsules containing ingestible sensors while wearing the Reader and being observed in a clinic setting.

ELIGIBILITY:
Stratification for gender and Body Mass Index is performed.

The BMI-Gender categories will be: Normal/Underweight (BMI<25), Overweight (BMI 25.0 to <30), and Obese (BMI>30.0); and Male/Female.

Inclusion Criteria:

* Men and women 18 years of age or older.

  * Enroll at least one subject and less than four subjects 65 years of age or older
  * Enroll at least one subject and less than four subjects 18 to 21 years of age
* For females of childbearing potential, negative urine pregnancy test at time of entry and assurance that a medically-accepted means of contraception will be used for the duration of the study. Able and willing to provide informed consent.
* Willing to adhere to all protocol requirements and study procedures.
* Adequate organ function at screening (defined for investigator in protocol)

Exclusion Criteria:

* Unable to take oral medications.
* Women who are pregnant, breast-feeding, or plan to become pregnant during the study, and females of childbearing potential who are not using a medically-accepted means of contraception.
* Medical condition which may affect passage through the gastrointestinal tract
* Known hypersensitivity to any component of the ingestible ID-Capsule
* Significant medical condition, psychiatric condition, current alcohol or drug abuse, or other condition which may preclude the study participant from being able to follow study procedures or to safely participate in the opinion of the investigator..
* Participation in an investigational product study (e.g., medical device or drug study) within 30 days prior to screening, or prior participation in an Ingestion Event Marker study.
* Presence of an active implantable electronic medical device.
* Positive screen for drugs of abuse (detection of drug for which a valid prescription exists is not exclusionary)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Gender at birth
Enrollment: 36 (Actual)
Dates: Start 2018-03-22 (Actual); Primary Completion 2018-05-01 (Actual); Study Completion 2018-06-01 (Actual)

PRIMARY OUTCOMES:
Positive Detection Accuracy (PDA) | Up to 10 days
  The number of active ingestible sensors detected divided by the number of active ingestible sensors administered under direct observation.
Negative Detection Accuracy (NDA) | Up to 10 days
  The number of inactive empty capsules not detected divided by the number of inactive empty capsules administered under direct observation. Determination of NDA will also include the number of monitoring periods with no ingestion events detected by the Reader divided by the number of specific monitoring periods performed for the purpose of detecting false positives.

SECONDARY OUTCOMES:
Number of Study Participants with Adverse Events as a Measure of Safety and Tolerability | Up to 10 days during ingestion events through the follow-up assessment scheduled within 3 to 5 days of the last ingestion
  Incidence of mild, moderate, and severe adverse events overall and related to the device; discontinuations due to adverse events

OTHER OUTCOMES:
Gender/BMI Effects | Up to 10 Days
  Effect of gender/BMI on the positive detection accuracy (covariate analysis) and other device performance measures
Detection time | Up to 60 minutes post ingestion
  Time from ingestion of ID-Capsule to first detection by the ID-Cap Reader
Signal Duration | Up to 90 minutes post ingestion
  Time from first to last detection of the signal from the ingested sensor by the ID-Cap Reader

CONTACTS AND LOCATIONS:
Overall Officials: Gary Connor, RN, Study Director — EtectRX, Inc.
Locations (1):
- Quotient Sciences, Jacksonville, Florida, United States

IPD SHARING:
Plan to Share IPD: No